CLINICAL TRIAL: NCT05166733
Title: A Retrospective Study of Reco Thrombectomy Stent for Intravascular Treatment of Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PengYa (Other)
Collaborators: Jingjiang People's Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); The Second Hospital of Nanjing Medical University (Other); Northern Jiangsu People's Hospital (Other); Yixing People's Hospital (Other)
Responsible Party: Sponsor-Investigator, PengYa, Principal Investigator, The First People's Hospital of Changzhou
Organization: The First People's Hospital of Changzhou (Other)
Other Study IDs: 2021（ke）CL274
Record Dates: First submitted 2021-12-02; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Neurology; Interventional Therapy
Keywords: ischemic stroke; Reco; endovascular treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the differences in the green channel process of stroke in various regions of the same province, to target and shorten the time delay of emergency process, and to explore the key technologies of endovascular treatment of acute ischemic stroke. To investigate the use and embolectomy effect of Reco, the first embolectomy stent in China, in economically developed areas. Health economic assessment (cost-benefit analysis) of ischemic stroke patients in various regions of the province.

DETAILED DESCRIPTION:
The Reco Embolectomy Stent is indicated for patients who cannot be treated with intravenous tissue activator (IVt-PA) or who have failed IVt-PA therapy and is intended to remove thrombus from a large intracranial vessel in patients with ischemic stroke to restore blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years
* The clinical diagnosis was acute ischemic stroke
* Large vascular lesions were detected by head CT, CTA, MRI, MRA or DSA
* Preoperative baseline NIHSS score > 4
* MRS 0-1 before this stroke
* Mechanical thrombectomy was performed
* Use Reco thrombectomy bracket

Exclusion Criteria:

* epileptic seizure
* Sudden coma
* Neurological loss symptoms quickly improved
* Imaging was negative, but clinical symptoms did not rule out subarachnoid hemorrhage
* Previous intracranial hemorrhage, subarachnoid hemorrhage, and brain tumor (with mass effect)
* History of head trauma within 3 months prior to surgery
* History of arterial puncture with difficulty in compression and hemostasis within one week prior to surgery
* Physical examination revealed evidence of active bleeding or trauma (e.g. fracture)
* Women are known to be pregnant or breastfeeding
* Severe allergies to contrast agents are known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endovascular treatment for acute ischemic stroke with the Reco Embolectomy Stent from December 2018 to June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The time between the onset of the disease and the opening of the blood vessels | Immediately after surgery
  Calculate the time from onset to vessel opening
Functional independence at 90 days (defined as mRS≤2) | 90day after surgery
  mRS scores were performed 90 days after surgery
Symptomatic intracranial hemorrhage within 24 hours after surgery | 24 hours after surgery
  Symptomatic intracranial hemorrhage was evaluated by CT 24 hours after operation

SECONDARY OUTCOMES:
Time from onset to admission | Immediately after surgery
  Calculate the time from onset to admission
Time from admission and puncture time | Immediately after surgery
  Calculate the time from onset to admission
Puncture to the time of vessel opening | Immediately after surgery
  Calculate the time from puncture to vascular opening

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No